CLINICAL TRIAL: NCT02246738
Title: Initial Evaluation of a Telomerase-based Circulating Tumor Cell Assay in Bladder Cancer Cohorts
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 07814
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Urothelial Carcinoma of the Bladder
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Collection
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- Cohort1
  Interventions: Other: Blood Collection
- Cohort 2
  Interventions: Other: Blood Collection
- Cohort 3
  Interventions: Other: Blood Collection
- Cohort 4
  Interventions: Other: Blood Collection
- Cohort 5
  Interventions: Other: Blood Collection
- Cohort 6
  Interventions: Other: Blood Collection
- Cohort 7
  Interventions: Other: Blood Collection
- Cohort 8
  Interventions: Other: Blood Collection
- Cohort 9
  Interventions: Other: Blood Collection

INTERVENTIONS:
Other: Blood Collection

SUMMARY:
Purposes are to determine whether various cohorts of bladder cancer patients have detectable tCTC's, determine it tCTC levels vary with the natural history of bladder cancer and to see if tCTC's provide novel information.Study population are various cohorts of patients diangosed with urothelial carcinoma of the bladder.Procedures include a venous blood draw, up to two times, over a 6 month period for collection of tCTC's. Up to 15 mL's of blood will be collected at each blood draw.

ELIGIBILITY:
Inclusion Criteria:

* a.Urothelial carcinoma or mixed urothelial carcinoma arising from the bladder
* b.Age 18 or older
* Inclusions by cohort Cohort 1. Patients with localized muscle-invasive disease (cT1,cN0, M0) at the time of initial diagnosis or who have progressed from superficial disease (cT2) who have not had any systemic chemotherapy and who will be treated with upfront radical cystectomy. PriorTURBT and intravesical therapies are allowed but should not have been done within one week of CTC measurement. If the patient is found to have no evidence of tumor (pT0) upon evaluation of the cystectomy specimen, the patient will not be dropped. If the patient is found to have evidence of progression by any clinical evaluation performed within 2 months of the post-treatment sample, the patient will be dropped from Cohort 1 and included in Cohort 9 instead.
* Cohort 2. Patients with localized muscle-invasive disease (cT1, cN0, M0) at the time of initial diagnosis prior to definitivechemo-radiation. Prior TURBT and intravesical therapies are allowed but should not have been done within one week of CTC measurement. If the patient is found to have evidence of progression by anyclinical evaluation performed within 2 months of the post-treatment sample, the patient will be droppedfrom Cohort 2 and included in Cohort 9 instead.
* Cohort 3. Patients with localized muscle-invasive disease (cT1, cN0, M0) at the time of initial diagnosis or who have progressed from superficial disease (cT2) who have not had any systemic chemotherapy and who will be treated with neoadjuvant chemotherapy. Prior TURBT and intravesical therapies are allowed but should not have been done within one week of CTC measurement. If the patient is found to have evidence of progression by any clinical evaluation performed within 2 months of the post-treatment sample, the patient will be dropped from Cohort 3 and included in Cohort 9 instead.
* Cohort 4. Patients with metastatic disease (anyT, anyN, M1) at initial presentation or recurrent after definitive treatment prior to any salvage systemic chemotherapy. If the patient is found to have evidence of progression by any clinical evaluation performed within 2 months of the post-treatment sample, the patient will be dropped from Cohort 4 and included in Cohort 9 instead.
* Cohort 5. Patients with newly diagnosed non-muscle-invasive bladder cancer (T2) prior to any intravesical therapy. If the patient is found to have evidence of progression by any clinical evaluation performed within 2 months of the post-treatment sample, the patient will be dropped.
* Cohort 6. Patients with muscle-invasive bladder cancer after radical cystectomy with or without peri-operative systemic chemotherapy (pT2, anyN, M0) who will be treated with adjuvant radiation. If the patient is found to have evidence of progression by any clinical evaluation performed within 2 months of the post-treatment sample, the patient will be dropped from Cohort 6 and includedin Cohort 9 instead.
* Cohort 7. Patients with a history of muscle invasive bladder cancer (cT1, any N,M0) who have no evidence of disease at least 2 years after the date of radical cystectomy. If the patient is found to have evidence of progression by any clinical evaluation performed within 2 months of the post-treatment sample, the patient will be dropped from Cohort 7 but may be considered for inclusion in Cohort 4.
* Cohort 8. Patients with a history of muscle invasive bladder cancer (cT1, any N, M0) who have no evidence of disease at least 2 years after the completion of definitive chemo-radiation. If the patient is found to have evidence of progression by any clinical evaluation performed within 2 months of the post-treatment sample, the patient will be dropped from Cohort 8 but may be considered for inclusion in Cohort 4.
* Cohort 9. Patients who were initially included in Cohorts 1-6 but were found to have progression at the time of their post-treatment blood draw. Of note, patients may be included in more than one cohort over time so long as inclusion and exclusion criteria are met. In addition, twenty samples from normal controls without any history of malignancy will be used for this study but havealready been collected as part of a separate protocol.

Exclusion Criteria:

* pure squamous or pure adenocarcinoma bladder cancer histology. This exclusion may be waved at the discretion of the protocol PI. 2. Prior cancer diagnosed within 3 years of enrollment other than a prior bladder, prostate, or skin cancer. This exclusion may be waved at the discretion of the protocol PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urothelial Carcinoma of the Bladder
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: John Christodouleas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States